CLINICAL TRIAL: NCT03318289
Title: Exercise is Medicine and Community Wellness - A Ving Tsun Martial Exercise Programme for Community-dwelling Older Adults
Brief Title: Ving Tsun Martial Exercise for Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1602061
Record Dates: First submitted 2017-10-09; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Old Age; Atrophy
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ving Tsun (VT) group (Experimental): Participants in the VT group will receive VT exercise intervention for 12 weeks.
  Interventions: Behavioral: Ving Tsun
- Control group (No Intervention): No intervention but can continue daily activities.

INTERVENTIONS:
Behavioral: Ving Tsun — The VT training regimen is designed to improve reactive balance control, lower extremity muscle strength and balance confidence in the elderly. It comprises 9 VT sticking-hand drills that must be practised with a partner. Participants will be trained to respond rapidly to upper body perturbations and to maintain body balance. Those joined the VT training group will attend a one-hour supervised VT training session at an elderly community centre 2 times per week for 12 weeks.
  Arms: Ving Tsun (VT) group

SUMMARY:
Objectives: To evaluate the effects of a Ving Tsun (VT) reactive balance training programme on reactive balance control, muscle strength, balance confidence and falls in community-dwelling older adults.

Hypothesis: The VT group subjects will have improved post-training reactive balance control, muscle strength, balance confidence and fall incidence outcomes than the active controls.

Design and subjects: In this prospective, randomised, single-blinded controlled trial, approximately 114 healthy seniors (55-70 years old) will be randomly assigned to either the VT group (n~57) or control group (n~57). Interventions: Subjects in the VT group will receive VT reactive balance training (3 hours/week) for 3 months, whereas subjects in the control group will receive no VT training but will jog 3 hours/week during the intervention period.

Study instruments and outcomes: Primary outcome measures: reactive balance control, as indicated by lower extremity muscle activation onset latency; hip and ankle strategies and centre of pressure movements will be measured by electromyography, electrogoniometry and a force platform, respectively. Secondary outcome measures: knee muscle strength, balance confidence and fall history will be assessed by an isokinetic dynamometer, Activities-specific Balance Confidence Scale (Chinese) and interviews, respectively (pre-, post- and follow-up measurements).

Data analysis: Data will be analysed using repeated-measures analysis of (co)variance followed by post-hoc tests, as appropriate (alpha = 0.05).

DETAILED DESCRIPTION:
Objectives:

To evaluate the effects of a Ving Tsun (VT) martial exercise programme on reactive balance control, lower limb muscle strength, balance confidence and falls in community-dwelling older adults.

Study design:

This will be a prospective, non-randomised and controlled intervention trial.

Subjects:

Approximately 40 healthy older adults will be recruited from elderly community centres by convenience sampling through poster advertising. Eligible subjects will be allocated to either the VT group (n ≈ 20) or control group (n ≈ 20).

Outcome measurements:

All subjects will be assessed before the intervention (baseline tests) and shortly after the 3-month intervention (post-tests). All subjects, regardless of group assignment, will undergo the following baseline tests and post-tests in random order.

Primary outcome measures Reactive balance control including lower extremity muscle activation onset latency and centre of pressure movement in standing.

Secondary outcome measures Lower extremity (knee) muscle strength, balance confidence and fall history.

Data analysis:

Data will be analysed using repeated-measures analysis of (co)variance followed by post-hoc tests, as appropriate (alpha = 0.05).

ELIGIBILITY:
Inclusion Criteria:

1. aged between 55 and 70 years,
2. able to ambulate independently,
3. an Abbreviated Mental Test (Hong Kong version) score > 7 and
4. able to follow commands and communicate with others.

Exclusion Criteria:

1. unstable medical condition (e.g. uncontrolled hypertension),
2. recent injury that may affect test performance,
3. history of fragility fractures,
4. significant musculoskeletal disorder (e.g. frozen shoulder),
5. sensorimotor disorder that may affect balance performance,
6. significant neurological disorder (e.g. stroke),
7. cardiopulmonary disease (e.g. chronic obstructive pulmonary disease),
8. cognitive disorders,
9. regular engagement in sports or martial arts training (e.g. Tai Chi) and
10. too frail to participate in VT intervention.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2020-10-09 (Estimated); Study Completion 2020-10-09 (Estimated)

PRIMARY OUTCOMES:
Lower extremity muscle activation onset latency | 3 months
  Lower extremity muscle activation onset latency in response to postural preturbation will be measured using surface electromyography.
Centre of pressure movement in standing | 3 months
  Centre of pressure movement in standing will be measured using a force platform.

SECONDARY OUTCOMES:
Knee maximum muscle strength | 3 months
  Knee maximum muscle strength will be measured by an isokinetic dynamometer.
Balance confidence | 3 months
  Balance confidence will be evaluated using the Activities-specific Balance Confidence Scale. Participants will be asked to rate on an 11-point scale ranging from 0 (no balance confident) to 100 (completely confident) for completing 16 daily activities while maintaining body balance. The mean of the total item score (0-100) will be used for analysis. Higher scores indicate better balance confidence.
Fall history | 3 months
  The number of falls and fall related injuries will be obtained through interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Fong, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fong SSM, Chung LMY, Yam TTT, Chung JWY, Bae YH, Gao Y, Chan JSM, Wang HK. Effects of Ving Tsun sticking-hand training on lower limb sensorimotor performance among community-dwelling middle-aged and older adults: a randomized controlled trial. Trials. 2023 Feb 25;24(1):143. doi: 10.1186/s13063-023-07133-2. PMID 36841770